CLINICAL TRIAL: NCT03515720
Title: Effectiveness of Neuroprolotherapy With Home Physical Therapy Against Isolated Physical Therapy for the Treatment of Patellar Chondromalacia
Brief Title: Neuroprolotherapy With Physical Therapy for Treatment of Patellar Chondromalacia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Full time surgical researcher, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Neuroproloterapia_2018
Record Dates: First submitted 2018-04-23; First posted 2018-05-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Chondromalacia Patellae
MeSH Terms: conditions — Chondromalacia Patellae | interventions — Prolotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Painful points will be located in the path of the sensory nerves of the knee in which asepsis and antisepsis will be performed, and then 0.5-1 ml of 5% dextrose solution will be applied subcutaneously at a 45º angle along the way. of the nerve with a 27 gauge needle of ½ inch. The number of injections will vary according to the symptoms to be treated. The application will be made once a week for 6 weeks. After the first application of neuroprolotherapy, the patient will be trained to perform a rehabilitation therapy program based on thermotherapy, kinesitherapy and knee strengthening exercises. At the end of the 6 sessions, a new assessment will be made with the WOMAC, EVA and measurement of movement arcs to assess the evolution after treatment.
  Interventions: Procedure: Prolotherapy
- Control group (No Intervention): Physical therapy consisting of 10 sessions based on thermotherapy, kinesitherapy and muscle strengthening exercises to the knee. Subsequently, the patient will perform this therapy home until completing 6 weeks. At the end a new assessment will be made with measurement of movement arcs, WOMAC scale and EVA to assess the evolution after treatment.

INTERVENTIONS:
Procedure: Prolotherapy — It consists of injecting 5% dextrose in sterile aqueous solution without the use of lidocaine in a subcutaneous nerve to inhibit neurogenic inflammation and the release of substance P and CGRP, decreasing neurogenic inflammation.
  Other Names: Neural prolotherapy
  Arms: Study group

SUMMARY:
Patellar chondromalacia is the degeneration of articular cartilage located on the posterior face of the patella and may suggest the onset of an osteoarthrosis. It predominates in sedentary people who overload the joint, as well as people with insufficiency in the extensor muscles of the knee. It is often seen between 30 and 40 years. Conservative management is the main treatment option and surgical intervention is considered as a last option in a small number of patients. A new treatment option is neuroprolotherapy where the approach is directed at the subcutaneous nerves as the source of pathology, which can lead to neurogenic inflammation and pain.

DETAILED DESCRIPTION:
Introduction: Patellar chondromalacia is the degeneration of articular cartilage located on the posterior face of the patella and may suggest the onset of an osteoarthrosis. It predominates in sedentary people who overload the joint, as well as people with insufficiency in the extensor muscles of the knee. It is often seen between 30 and 40 years. Conservative management is the main treatment option and surgical intervention is considered as a last option in a small number of patients. A new treatment option is neuroprolotherapy where the approach is directed at the subcutaneous nerves as the source of pathology, which can lead to neurogenic inflammation and pain.

Objective: To evaluate the efficacy of neuroprolotherapy combined with a home physical therapy program in patients with a diagnosis of patellar chondromalacia against a control group receiving only physical therapy at home.

Methodology: Randomized clinical trial. We studied patients from the Rehabilitation Service with clinical and radiographic diagnosis of patellar chondromalacia. Two groups were studied: the first group received treatment with neuroprolotherapy combined with home physical therapy and the second group was managed with physical therapy alone, measuring the results by the WOMAC test at baseline and at 6 weeks thereafter.

Statistic analysis: The statistical analysis will be carried out in two stages, descriptive and analytical. In the first, the variables are presented as raw numbers, proportions and means of central tendency and dispersion. The analytical stage between the groups will be done by means of the Chi square test, or Fisher's exact test if any of the values of the tetra-table is equal or less than 5, for qualitative variables. For the quantitative variables an analysis of equality of variance of Levene will be made, and if the results have a normal behavior, the Student's T test will be performed, otherwise it will be analyzed with the Man Withney U test. For the intra-group analysis, the response variables before and after the treatment assigned by randomization will be included, and for the analysis of the quantitative variables, the Student's T test for related samples and the Chi-square test or Fisher's Exact test will be used for the qualitative. Any P value less than 0.05 will be considered statistically significant. The results will be captured in a database in Excel for Windows. For the statistical analysis, the SPSS program for Windows version 23 will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in the rehabilitation medicine service of the Specialties Hospital National Medical Center of the West.
* Men and women with clinical and radiographic diagnosis of chondromalacia patellae with or without gonarthrosis.
* Age over 25 years
* Patients expressed their signed consent to participate in the study....

Exclusion Criteria:

* Patients who have been infiltrated with corticosteroids in the knee during the last year.
* Septic arthritis.
* Systemic infection or cutaneous infection at the site of infiltration.
* Systemic inflammatory disease.
* Joint instability (ligament injuries).
* Meniscopathies
* Intra-articular fracture
* Coagulation disorder or treatment with anticoagulants.
* Diabetes mellitus poorly controlled (> 130mg / dL).
* Badly controlled systemic arterial hypertension (> 140 / 90mmHg).
* Hemarthrosis
* Pregnancy.
* Patients with cognitive disorders that prevent the follow-up of indications or carry out the program.
* Patients who do not accept to sign informed consent.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
WOMAC Osteoarthritis Index | 6 weeks
  The WOMAC Osteoarthritis Index is a specific instrument for osteoarthrosis. It was developed to have a standard and internationally valid measuring instrument to evaluate the results in clinical trials of knee and hip osteoarthritis treatments preferably. It selects three important concepts for the patient and independent of the observer: pain, rigidity and functional capacity. The WOMAC Osteoarthritis Index is obtained from a questionnaire that uses a visual analogical scale for the evaluation of pain (6 questions), rigidity (2 questions) and physical function (17 questions). The best score for each item is 0, using an analog visual scale of 10 centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Cleotilde Fuentes Orozco, PhD, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Roberto Mares País, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Sandra Angélica García Triana, MD, Principal Investigator — Unit of Physical Medicine and Rehabilitation, High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; María Fernanda Toro Sashida, MD, Principal Investigator — Unit of Physical Medicine and Rehabilitation, High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute; Francisco José Barbosa Camacho, MD, Principal Investigator — High Specialty Medical Unit, National Western Medical Center, Mexican Social Security Institute
Locations (1):
- Centro Médico Nacional de Occidente, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YM, Joo YB. Patellofemoral osteoarthritis. Knee Surg Relat Res. 2012 Dec;24(4):193-200. doi: 10.5792/ksrr.2012.24.4.193. Epub 2012 Nov 29. PMID 23269956
- [Background] Weglein A. Neural prolotherapy Wonder Why? Journal of Prolotherapy. May 2011; 3(2): 639-643.
- [Background] Hauser R, Maddela H, Alderman D, Baehnisch G, Banner R, Blakemore P et al. Journal of Prolotherapy International Medical Editorial Board Consensus Statement on the Use of Prolotherapy for Musculoskeletal Pain. Dec 2011;3(4):744.
- [Background] Reeves KD, Hassanein K. Randomized prospective double-blind placebo-controlled study of dextrose prolotherapy for knee osteoarthritis with or without ACL laxity. Altern Ther Health Med. 2000 Mar;6(2):68-74, 77-80. PMID 10710805
- [Background] Hauser RA, Sprague IS. Outcomes of prolotherapy in chondromalacia patella patients: improvements in pain level and function. Clin Med Insights Arthritis Musculoskelet Disord. 2014 Feb 17;7:13-20. doi: 10.4137/CMAMD.S13098. eCollection 2014. PMID 24596471
- [Background] Haspl M, Dubravcic-Simunjak S, Bojanic I, Pecina M. [Anterior knee pain associated with sports and work]. Arh Hig Rada Toksikol. 2001 Dec;52(4):441-9. Croatian. PMID 11831127
- [Background] Rezasoltani Z, Taheri M, Mofrad MK, Mohajerani SA. Periarticular dextrose prolotherapy instead of intra-articular injection for pain and functional improvement in knee osteoarthritis. J Pain Res. 2017 May 17;10:1179-1187. doi: 10.2147/JPR.S127633. eCollection 2017. PMID 28553139
- [Result] Maniquis-Smigel L, Dean Reeves K, Jeffrey Rosen H, Lyftogt J, Graham-Coleman C, Cheng AL, Rabago D. Short Term Analgesic Effects of 5% Dextrose Epidural Injections for Chronic Low Back Pain: A Randomized Controlled Trial. Anesth Pain Med. 2016 Dec 6;7(1):e42550. doi: 10.5812/aapm.42550. eCollection 2017 Feb. PMID 28920043
- [Result] Yelland MJ, Sweeting KR, Lyftogt JA, Ng SK, Scuffham PA, Evans KA. Prolotherapy injections and eccentric loading exercises for painful Achilles tendinosis: a randomised trial. Br J Sports Med. 2011 Apr;45(5):421-8. doi: 10.1136/bjsm.2009.057968. Epub 2009 Jun 22. PMID 19549615
- [Result] Jara-Oseguera A, Simon SA, Rosenbaum T. TRPV1: on the road to pain relief. Curr Mol Pharmacol. 2008 Nov;1(3):255-69. doi: 10.2174/1874467210801030255. PMID 20021438
- [Result] Fulkerson JP, Arendt EA. Anterior knee pain in females. Clin Orthop Relat Res. 2000 Mar;(372):69-73. doi: 10.1097/00003086-200003000-00009. PMID 10738416
- [Result] Friedman AH. An eclectic review of the history of peripheral nerve surgery. Neurosurgery. 2009 Oct;65(4 Suppl):A3-8. doi: 10.1227/01.NEU.0000346252.53722.D3. PMID 19927076
- [Result] Rabago D, Zgierska A, Fortney L, Kijowski R, Mundt M, Ryan M, Grettie J, Patterson JJ. Hypertonic dextrose injections (prolotherapy) for knee osteoarthritis: results of a single-arm uncontrolled study with 1-year follow-up. J Altern Complement Med. 2012 Apr;18(4):408-14. doi: 10.1089/acm.2011.0030. PMID 22515800
- [Derived] Garcia-Triana SA, Toro-Sashida MF, Larios-Gonzalez XV, Fuentes-Orozco C, Mares-Pais R, Barbosa-Camacho FJ, Guzman-Ramirez BG, Pintor-Belmontes KJ, Rodriguez-Navarro D, Brancaccio-Perez IV, Esparza-Estrada I, Bernal-Hernandez A, Gonzalez-Ojeda A. The Benefit of Perineural Injection Treatment with Dextrose for Treatment of Chondromalacia Patella in Participants Receiving Home Physical Therapy: A Pilot Randomized Clinical Trial. J Altern Complement Med. 2021 Jan;27(1):38-44. doi: 10.1089/acm.2020.0287. Epub 2020 Nov 20. PMID 33217236